CLINICAL TRIAL: NCT05559021
Title: What Concept of Manual Therapy is More Effective to Improved Health Status in Women With Fibromyalgia Syndrome?: An Experimental Study
Brief Title: What Concept of Manual Therapy is More Effective?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Eleuterio Atanasio Sánchez Romero, Principal Investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Concept of Manual Therapy
Record Dates: First submitted 2022-09-22; First posted 2022-09-29 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Quality of Life; Self Efficacy; Kinesiophobia; Catastrophizing; Central Sensitisation; Anxiety; Depression; Sleep
Keywords: Manual Therapy; Chronic Pain; Fibromyalgia; Passive Mobilizations; Myofascial Approach; Symptom Severity
MeSH Terms: conditions — Kinesiophobia; Anxiety Disorders; Depression; Chronic Pain; Fibromyalgia

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be conducted between October 2022 and December 2023 in 52 female patients impacted by Fibromyalgia who will undergo a myofascial treatment approach or mobilization treatment approach , with 3 months of follow-up post-treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Treatment Approach (Experimental): Patients will have 1 session per week, during 4 weeks, making 4 sessions in total. Each session will last 30 minutes. Each session consists of:
  * Transverse planes in the thoracolumbar fascia and abdomen: The physical therapist place his hands facing each other so that one hand is between the tables and the patient's thoracolumbar fascia and the other on the abdomen
  * Transverse planes at C7-D3 and sternum: The physical therapist, places one hand between the table and the patient's first 4 thoracic vertebrae (C7-T4) and the other on the sternum.
  * Suboccipital inhibition: the physical therapist, places his hands under the patient's head transversely between the occipital and the spinous process of C2. After, the head is lowered in such a way that the occipital bone rests on the tenar eminences and a slight traction is maintained cranially.
  Interventions: Other: Myofascial Therapy Treatments
- Mobilization Approach. (Experimental): Patients will have 1 session per week, for 4 weeks, which means 4 sessions in total. Each session will last 30 minutes. Each session consists of:
  * Postero-anterior cervical sliding: the patient's cervical vertebrae will be evaluated with the 4 degrees of postero-anterior sliding, and the pain at each vertebral level is recorded. Then, the most painful vertebra previously detected will be treated.
  * Postero-anterior lumbar slippage: the patient's lumbar vertebrae will be evaluated with the 4 degrees of postero-anterior slippage, and the pain at each vertebral level is recorded. Afterwards, the most painful vertebra previously detected will be treated.
  * Postero-anterior dorsal slippage: the patient's dorsal vertebrae will be evaluated with the 4 degrees of postero-anterior slippage, and the pain at each vertebral level is recorded. Then, Afterwards, it will treat during the most painful vertebra previously detected.
  Interventions: Other: Passive Mobilizations Approach

INTERVENTIONS:
Other: Myofascial Therapy Treatments — • Myofascial approach: After the bibliographic review of myofascial therapy treatments in fibromyalgia patients based on the articles by CastroSánchez AM et al., and an expert consensus, the following approach was decided: patients would have 4 sessions in total with 1 session per week of 30 minutes each.
  * Transverse planes in the thoracolumbar fascia (TCL) and abdomen: Performing a myofascial induction as described by Pilat.
  * Transverse planes at C7-D3 and sternum: Performing a myofascial induction as described by Pilat.
  * Suboccipital inhibition: Performing a myofascial induction as described by Pilat
  Arms: Myofascial Treatment Approach
Other: Passive Mobilizations Approach — • Approach with passive mobilizations: After the literature review of manual therapy treatments in fibromyalgia patients and a consensus of experts in Manual Therapy with more than 15 years of experience, the following approach was agreed upon by the expert: patients would have 4 sessions in total with 1 session per week of 30 minutes each.
  * Postero-anterior cervical sliding
  * Postero-anterior lumbar slippage
  * Postero anterior dorsal slippage
  Arms: Mobilization Approach.

SUMMARY:
The aim of the study will be to find out which manual therapy approach is most effective for the improvement of symptoms (sensory, cognitive, emotional and social) in people with Fibromyalgia.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted in 52 patients with Fibromyalgia who will undergo a myofascial treatment approach or a passive mobilization treatment approach. Data will be collected on the improvement of symptom severity, quality of life, self-efficacy, kinesiophobia, catastrophizing, central sensitization, anxiety, depression, and sleep. After the treatments, follow-ups will be made, and the results are expected to be disseminated to the scientific community during and after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Less than 62 years old
* Medical Diagnosis of Fibromyalgia
* The individuals included in the study had a minimum one-year history of symptoms
* To confirm the medical diagnosis of fibromyalgia, the physical therapists and study investigators used the 2010 American College of Rheumatology (ACR) diagnostic criteria. -Since 2 of the measurement variables used in the study (WPI and SS-Score) match the protocol when determining these criteria, this procedure was facilitated.

The diagnostic criteria establish the diagnosis of fibromyalgia when12 : IDG/WPI ≥ 7 and SS ≥ 5 or IDG/WPI 4-6 and SS ≥ 9.

Exclusion Criteria:

* Intolerance to touch
* A change of medication in the last 2-3 months
* Agree not to change their medication during the study

Exclusion Criteria:

-

Ages: 18 Years to 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — An experimental study will be conducted at the Fibromyalgia and Chronic Fatigue Association of Móstoles, Madrid, Spain. This is an all-female center. However, the prevalence of fibromyalgia is much higher in women (5:1 ratio, with respect to men), so the next study is highly relevant.
Enrollment: 52 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Pain Expansion | Change from baseline, immediately after the intervention with the different manual therapy protocols; and at 1, 2 and 3 months of follow-up after intervention
  This will be classified as a continuous numerical variable measured by the Widespread Pain Index (WPI). In this index, the patient has to mark with an x the areas in which he/she has presented pain during the last week
Symptom severity | Change from baseline, immediately after the intervention with the different manual therapy protocols; and at 1, 2 and 3 months of follow-up after intervention
  This variable will be classified as a continuous numerical variable, measured by the Symptom Severity Index (SSI/SS-Score), composed of two subscales (SS-1 and SS-2) that assess the intensity during the last week of 3 of the main symptoms present in FM (fatigue, unrefreshing sleep and cognitive disorders), as well as the presence/absence of other common symptoms, respectively. The total score of the SSS is the sum total and ranges from 0 to 12. The SSS correlated correlates strongly with the WPI (r=0.733) and with the presence of Tender Points (r=0.680)
Fibromyalgia Impact Questionnaire | Change from baseline, immediately after the intervention with the different manual therapy protocols; and at 1, 2 and 3 months of follow-up after intervention
  Another measurement variable will be the impact of fibromyalgia on quality of life, through the Fibromyalgia Impact Questionnaire (FIQ), a tool translated into Spanish by means of the international translation-retrotranslation recommendations, and whose reliability, validity, adaptation and sensitivity to change have been satisfactorily analyzed in Spanish patients with fibromyalgia. Consists of 19 items that measure three main categories (a) "function" - ten items that as-sess the participant's physical functions that address the participant's ability to perform each activity. This domain is assessed on a 4-point Likert scale, from 0 to 3 (0= always, 1= always, 1= always, 2= always, 3= always). 0 to 3 (0= always, 1= frequently, 2= occasional-ly, 3= never). (b) "Global impact" - composed of two items assessing the number of days in the last week when the participants felt good and the number of days they could not work due to FM symptoms

SECONDARY OUTCOMES:
kinesiophobia | Change from baseline, immediately after the intervention with the different manual therapy protocols; and at 1, 2 and 3 months of follow-up after intervention
  For this purpose, we will use the Tampa Kinesiophobia Scale (TSK), also translated and validated in Spanish. It is a 17-item self-report measure that will be used to measure fear of movement. A high score indicates an extreme fear of movement, while a low score indicates a negligible fear of movement.
Self-Efficacy | Change from baseline, immediately after the intervention with the different manual therapy protocols; and at 1, 2 and 3 months of follow-up after intervention
  For this purpose, we will use the Pain Self-Efficacy Questionnaire, in its Spanish validated version. The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire developed to assess the confidence that people with persistent pain have in performing activities while in pain. The PSEQ is applicable to all presentations of persistent pain. It inquires about the level of self-efficacy in relation to a range of functions, such as housework, socializing, work, as well as coping with pain without medication. The PSEQ is a 10-item questionnaire developed to assess the confidence that people with persistent pain have in performing activities while in pain. The PSEQ is applicable to all presentations of persistent pain. It inquiries about the level of self-efficacy in relation to a range of functions, such as housework, socializing, work, as well as coping with pain without medication.
Anxiety | Change from baseline, immediately after the intervention with the different manual therapy protocols; and at 1, 2 and 3 months of follow-up after intervention
  The the State-Trait Anxiety Inventory (STAI) questionnaire will be used to assess two independent concepts of anxiety, each with 20 items:
  Anxiety as a state: assesses a transient emotional state, characterized by subjective, consciously perceived feelings of alertness and apprehension and by hyperactivity of the autonomic nervous system.
  Anxiety as a trait: indicates a relatively stable anxious propensity that characterizes individuals with a tendency to perceive situations as threatening.
Depression | Change from baseline, immediately after the intervention with the different manual therapy protocols; and at 1, 2 and 3 months of follow-up after intervention
  The Beck Depression Inventory is a useful tool to assess somatic symptoms of depression, both in anxiety disorders and depressive conditions. The questionnaire consists of 21 questions, providing a range of scores between 0 and 63.
  The questionnaire proposes the following cut-off scores and corresponding degrees of depression: 0-13 indicates minimal depression, 14-19 mild depression, 20-28 moderate depression and 29-63 severe depression.
Quality of life (EQ-5D-5L) | Change from baseline, immediately after the intervention with the different manual therapy protocols; and at 1, 2 and 3 months of follow-up after intervention
  It will be evaluated by means of the the EuroQol 5-dimensions 5-levels (EQ-5D-5L), which is a generic instrument for measuring health-related quality of life. The patient himself assesses his state of health, in levels of severity by dimensions The first allows the respondent to define the state of health according to the EQ-5D multi-attribute classification system, composed of 5 dimensions (mobility, self-care, activities of daily living, pain/discomfort and anxiety/depression), and in each of them there are 3 levels of severity (1, 2 or 3).
Sleep quality | Change from baseline, immediately after the intervention with the different manual therapy protocols; and at 1, 2 and 3 months of follow-up after intervention
  The Pittsburgh Sleep Quality Index (PSQI) consists of 19 self-administered questions and 5 questions assessed by the patient's partner or roommate (if available). Only the self-administered questions are included in the score.
  The PSQI, developed by the Department of Psychiatry at the University of Pittsburgh in 1988, is a questionnaire that assesses both qualitative and quantitative aspects of sleep quality in the month prior to its administration.
  It shows that subjective sleep quality, duration, efficiency, disturbances and daytime dysfunction have better quality in those with moderate and severe impairment; while in those with average and higher performance, higher sleep latencies are observed. The total score is 21, and scores above 5 indicate significant sleep disturbance.
Visual Analog Scale (VAS) | Change from baseline, immediately after the intervention with the different manual therapy protocols; and at 1, 2 and 3 months of follow-up after intervention
  To evaluate the pain that the patient has, we use the VAS. This is a 100 mm line that measures pain intensity. The left end of the line represents the absence of pain, while the right end represents the worst pain imaginable. The numerical pain intensity scale adds a numerical graduation where 1 is no pain and 10 is the worst pain imaginable. The confidence and reliability of this scale has been approved and validated in different studies.

CONTACTS AND LOCATIONS:
Overall Officials: Eleuterio A. Sánchez Romero, PhD, Principal Investigator — European University of Madrid
Locations (2):
- Spain (2):
  - Eleuterio A. Sánchez Romero, Madrid
  - Universidad Europea de Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No